CLINICAL TRIAL: NCT03886818
Title: Evaluation of the Efficacy of Negative Pressure Wound Therapy on Incisional Wound Healing After a Total Ankle Arthroplasty: a Randomized Study.
Brief Title: Efficacy of Negative Pressure Wound Therapy After Total Ankle Arthroplasty
Acronym: PICO-PTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL18_0753
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Ankle Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICO strategy (Experimental): * Use of PICO™ device from the ankle surgery to the post-surgery day 7.
  * Use of usual care by simple dressings after post-surgery day 7 up to wound healing
  Interventions: Device: PICO strategy
- Standard of care (Active Comparator): -Usual care by simple dressings after the ankle surgery until the wound healing.
  Interventions: Device: Standard dressings

INTERVENTIONS:
Device: Standard dressings — Standard dressings will be used from surgery to wound healing
  Arms: Standard of care
Device: PICO strategy — The PICO system with negatif pression will be used from surgery to day 7. After that, standard dressing will be used untill the wound Healing.
  Arms: PICO strategy

SUMMARY:
About 500 total ankle prostheses are implanted each year in France. Wound healing issues are the most common complications after Total Ankle Arthroplasty (TAA). In 2010, a French retrospective study observed a wound infection rate of 8% among 592 prostheses implanted. Wound infection rate can vary up to 28% from the data available in the literature. Delayed wound healing is a known risk factor of surgical site infection (SSI). Even if it remains a rare event, its consequences for the patient can be severe and lead to removal and/or replacement of the prosthesis, arthrodesis, or transtibial amputation.

Negative Pressure Wound Therapy (NPWT) is an adjuvant therapy for wound management and healing: it delivers a controlled negative pressure (sub-atmospheric) applied topically onto the wound from a vacuum pump. The wound is filled with wound filler and sealed with an airtight adhesive drape. It allows creating a moist wound environment, removing exudate, and reducing edema and risk of infection.

Incisional NPWT can accelerate wound healing regardless of the surgery performed, including orthopedics. A retrospective study compared the incidence of healing complications after TAA between the administration of the NPWT PICO™ (Smith&Nephew) and the standard of care of postoperative wounds in 74 patients. A significant reduction of wound healing issues (3% vs. 24%, respectively; p=0.004) and a non-significant reduction of SSI (3% vs. 8%, respectively) were observed.

To the investigator knowledge, no randomized study has been conducted to assess the efficacy of the NPWT PICO™ for postoperative wound healing after TAA: Investigators propose to set up this study to obtain a high level of evidence in this population and investigators assume that the use of the PICO™ system after TAA would reduce delayed wound healing compared to the standard of care with conventional dressings.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Patient for whom a total ankle arthroplasty has been scheduled
* Patient affiliated to a national health insurance scheme or similar
* Patient who have signed an informed consent form for its participation in the study

Exclusion Criteria:

* Patient with contraindication to use of the PICO™ device
* Patient participating in another study including an exclusion period in progress
* Patient participating in another interventional study that may interfere with this research
* Adult patient protected by law, under guardianship or tutorship ;
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
Number of days from suture removal (i.e. day 21 after surgery) to achieve complete wound healing defined as: no visible exudate on protection dressing; and no blister; and no necrosis; and no wound dehiscence. | Up to 12 months after TAA

SECONDARY OUTCOMES:
Rate of technical failures of the PICO™ device, and type of failure: device failure, non-hermetic dressing, other. | baseline to postoperative day 7
Number and type of adverse effects related to the PICO™ device. | baseline to postoperative day 7
Rate of wound healing complications: presence of exudate; blister; necrosis; wound dehiscence. | postoperative day 21, postoperative week 6, postoperative months 4 and 12.
Rate of surgical site infection (superficial, deep or of a surgical site other than the incision site). | postoperative day 30 to postoperative month 12.
Rate of surgical revision for wound healing complications defined by: mechanical debridement; surgical debridement; flap surgery and skin graft. | Baseline to postoperative month 12.
Incremental Cost-Effectiveness Ratio (ICER) between the two dressing strategies. | Up to 12 months after TAA.
  A cost-effectiveness analysis comparing the strategy using PICO device and the one using only conventional dressing will be performed during 12 months after surgery, from the perspectives of the French hospital and French health insurance system; the result will be expressed in terms of cost per complication avoided.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Dr BESSE, Principal Investigator — Hospice Civils de Lyon
Locations (1):
- Service de Chirurgie orthopédique - Groupement Hospitalier Lyon Sud, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided